CLINICAL TRIAL: NCT02880072
Title: Absorption of Orally Ingested Phosphate in Head and Neck Cancer Patients With and Without Refeeding Syndrome
Brief Title: Absorption of Orally Ingested Phosphate in Refeeding Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, MD, MPA, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-6-2013-001
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Refeeding Syndrome; Cancer of the Head and Neck
MeSH Terms: conditions — Refeeding Syndrome; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- refeeding syndrome (Experimental): 6 patients with head and neck cancer and refeeding syndrome, 4 different of preparations of phosphate orally
  Interventions: Dietary Supplement: phosphate orally
- no refeeding syndrome (Experimental): 6 patients with head and neck cancer without refeeding syndrome, 4 different of preparations of phosphate orally
  Interventions: Dietary Supplement: phosphate orally

INTERVENTIONS:
Dietary Supplement: phosphate orally — 4 different preparations of phosphate

SUMMARY:
A phosphate supplement is part of the treatment of patients with the refeeding syndrome (RFS). It is not known, if the generalized edema also affects the intestine to decrease absorption. The aim was to investigate, if oral treatment is possible in mild to moderate RFS. In a randomized crossover design 12 hospitalized head-neck cancer patients ingested four oral solutions of phosphate in two-day periods. In a low-dose period the investigators compared five mmol phosphate from either skimmed milk or Di-sodiumphosphate-di-hydrate and potassium di-hydrogens-phosphate with black currant flavor (PBC), and in a high-dose period 20 mmol from either Addiphos® or the PBC-solution. P-phosphate was measured two and four hours after the ingestion, the urinary excretion after four hours.

P-phosphate significantly increased after PBC in both the low- and high-dose and Addiphos®, but not after skimmed milk. The increase was larger after Addiphos® than the PBC-solution. There was no difference in the increase between the patients with low p-phosphate and those with normal values, and no correlation between baseline p-phosphate and percent increase. There was no group difference in the urinary excretion of phosphate. The investigators conclude that phosphate can be readily absorbed after oral administration, but skimmed milk can´t be recommend for this purpose.

DETAILED DESCRIPTION:
The study was designed as a non-blinded, randomized, controlled crossover intervention study.

A total of 12 hospitalized adult head-neck cancer patients, 11 men and one woman, gave informed consent to participate. Six patients with a p-phosphate between 0.30-0.80 mmol/l were included as well as six patients (controls) with a p-phosphate in the normal range of 0.80-1.50 mmol/l. The control patients matched the hypophosphatemic patients regarding sex, age (± 10 years) and alcohol habits. Patients with diagnosed renal failure, edema, diabetes, liver failure, gastrointestinal disorders, pregnant and lactating women were excluded. None of the patients had phosphate supplementation within the previous 24 h. Randomization determined the order of the phosphate supplements divided into low-doses of five mmol followed by high-dose 20 mmol both for two day periods. Accordingly, four days intervention with a different phosphate supplement every day.

In the low-dose period supplements consisted of a daily dose of five mmol phosphate from skimmed milk (97 mg phosphorus and 0.1 g fat/100 ml) or Phosphate with black currant flavor (PBC) (disodiumphosphatedihydrate and potassiumdihydrogenphosphate, 1 mmol phosphate/ml). In the high-dose period supplements consisted of 20 mmol phosphate from Addiphos® (Fresenius-Kabi) (disodiumphosphate, potassiumdihydrogenphosphate, potassiumhydroxide, 2 mmol/ml) and PBC. The patients fasted six hours prior to baseline blood- and urine samples and during the four hours of the trial. Blood samples were repeated after two and four hours, urine after four hours. The interval between blood samples was determined on the basis of an animal experiment, which described phosphate absorption measured in plasma 1 hour after administration (10). The interval was extended to 2 hours due to the risk of gastric retention.

The primary outcome was the changes in p-phosphate. The secondary outcomes were changes in u-phosphate and changes in p-potassium, p-magnesium and p-sodium. The paired data were tested by the Wilcoxon test. Non paired data were tested by the Mann-Whitney test. Spearman-rank correlation test was used, and the statistical analyses were performed with STATA version 13.1 (StataCorp LP, USA, Texas).

ELIGIBILITY:
Inclusion Criteria:

* Head and Neck cancer diagnosed + informed consent

Exclusion Criteria:

* Severe organ failure, pregnancy, lactating women, in treatment with phosphate, unable to communicate sufficiently to understand the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
plasma phosphate | 4 hours
  measurements up till 4 hours after oral ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, MD, MPA, Principal Investigator — University of Copenhagen
Locations (1):
- Clinic for Ear, Nose and Throat Surgery, Rigshospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No